CLINICAL TRIAL: NCT03663790
Title: Comparison of the Effects of Gait Modification Strategies on Knee Adduction Moment in Patients With Medial Knee Osteoarthritis: Randomized Controlled Trial
Brief Title: Effects of Gait Retraining on Lower Extremity Biomechanics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Gait retraining OA
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; biomechanics; gait retraining; real-time biofeedback; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Foot Progression (Experimental): Participants will visualize a desired foot progression angle bandwidth in real-time that they should target with their foot angle
  Interventions: Other: Foot Progression
- Trunk Lean (Experimental): Participants will visualize a desired trunk lean angle bandwidth in real-time that they should target with their trunk lean angle
  Interventions: Other: Trunk Lean

INTERVENTIONS:
Other: Foot Progression — The intervention will be a gait retraining biofeedback focused on foot angle during gait trials
  Arms: Foot Progression
Other: Trunk Lean — The intervention will be a gait retraining biofeedback focused on trunk lean angle during gait trials
  Arms: Trunk Lean

SUMMARY:
The purpose of this proposed study is to investigate both the acute and chronic response of frontal plane knee moment after gait retraining and to assess the effects on the biomechanics of the contralateral side. Fifty-one patients diagnosed with tibiofemoral joint osteoarthritis (TFJ OA) will be recruited to participate in the proposed study. Participants will complete baseline trials to assess gait kinematic and kinetic parameters. Following baseline, each participant will perform six conditions of the foot progression gait or three conditions of the trunk lean gait modifications to determine which strategy is most effective in reducing frontal plane knee moment. Participants will then be randomized to either the control or experimental group based on their identified preferred strategy.

Participants will complete eight gait retraining sessions using patient-specific gait modifications (tailored foot progression and tailored lateral trunk lean), or normal gait (control) during the training period. A fading feedback design will be implemented. Real-time haptic biofeedback will be provided on every step during the first two weeks and reduced by 25% every subsequent two weeks. No feedback will be provided during baseline and at testing sessions. Measures of pain and function will also be collected at all testing sessions. Variables of interest include ankle, knee, hip sagittal and frontal plane moments. In addition, sagittal and frontal plane impulse will also be assessed.

Descriptive statistics will be calculated for foot progression angle, trunk lean angle, frontal and sagittal plane hip, knee, and ankle angles as well as moments. Descriptive statistics for frontal plane knee impulse will also be calculated. A multivariate analysis of variance (MANOVA) will be conducted to compare frontal plane knee moment, frontal plane knee impulse and the absolute sagittal plane moment will be compared across three groups at four different time points. Repeated measures analysis of variance (ANOVA) will be conducted to compare both sagittal and frontal plane joint biomechanics for the contralateral limb. The p-value will be set at .05.

DETAILED DESCRIPTION:
A randomized controlled study design with a waitlist will be used to investigate the effects of a 10-week gait retraining intervention on the knee adduction moment. Participants will be randomly assigned to either the intervention group or the control group. The intervention group will be further split into two groups. One group will consist of participants who reduced knee adduction moment (KAM) most with altered foot progression gait and the other will consist of participants who reduce KAM most effectively with trunk lean gait during pre-assessment. Participants will then perform 8 gait retraining sessions over 8 weeks (one session per week) using either their specific gait modification strategy (intervention) or with their normal gait (control). As part of the waitlist design, at the end of 10 weeks, patients assigned to the control group will be reassigned to their previously determined patient specific gait modification intervention. The goal is to minimize attrition and to increase the effective sample size.

On arrival to the laboratory, participants will be required to read and sign an informed consent form. Participant height and mass will be recorded. Pain and function will be assessed using the Western Ontario and McMaster Universities Arthritis (WOMAC) questionnaire and a numeric rating scale (NRS) from zero to 10, where zero represents no pain and 10 the highest level of pain. The experimental limb for the purpose of this study is defined as the leg diagnosed with symptomatic TFJ OA or the most symptomatic limb in the case of bilateral OA. Participants will be equipped with 4 surface electromyogram (sEMG) placed on the rectus femoris, vastus medialis, bicep femoris and semitendinosus of the experimental limb. EMG sensors will be used to record muscle activity during the baseline test. Participants will then have 53 retroreflective markers attached to their trunk and lower extremities. A static calibration trial of the VICON motion capture system will be acquired by having the participants stand on the foremost force plate with both feet aligned with the anterior-posterior axis of the laboratory. Participants will also perform a dynamic calibration by completing three clockwise rotations of the hip which will be used to estimate the hip joint centers. Participants will then complete 5 baseline walking trials along with a 6-meter walkway at their preferred speed. Participants will be required to walk for 12 minutes on a treadmill, and additional data will be recorded. Participants will then be required perform 9 conditions with altered foot progression gait or trunk lean gait to determine which strategy is most effective in reducing KAM. Participants will first receive standardized verbal instructions on how to achieve the instructed gait modification. Participants will then be provided haptic real-time biofeedback to ensure that they successfully achieve the required magnitudes of gait modification. Kinematic data collected in Vicon will be streamed to Matlab (Mathworks, Natick, MA) for real-time computation of joint angles. Participants will receive feedback from tactile sensors attached either to the lateral-proximal aspect of the fibula (foot progression) or the center of the scapula (lateral trunk lean) of the experimental side with hypoallergenic double-sided tape. One vibration will indicate a required decrease in the target gait parameter, while two vibrations will indicate a required increase. Feedback will be provided on each step and no vibration will indicate that no correction is needed. A trial will only be considered valid if the participant fully contacted the force plates twice with the foot of the experimental limb and the modified parameter was in the prescribed target range. Additionally, participants will be required to maintain an average gait speed ±5% relative to baseline for trials to be considered successful. The modification to be completed in the baseline session will be randomized for each participant. Once these trials are completed, participants will return to the lab within the same week to complete 5 additional baseline trials and three trials of whichever gait modification they did not perform the first day. Each baseline data collection session will take approximately one hour.

Participants will then be randomly assigned to either the intervention group or the control group. The intervention group will be further split into two groups. One group will consist of participants who reduced KAM most with altered foot progression gait and the other will consist of participants who reduce KAM most effectively with trunk lean gait. Participants will then perform 8 gait retraining sessions over 8 weeks (one session per week) using either their specific gait modification strategy (intervention) or with their normal gait (control). During gait-retraining sessions, participants will walk on a Woodway Desmo treadmill (Woodway, Waukesha, WI) placed in the center of a calibrated volume area (approximately 0.5 x 1.5 meters). A three-camera high-speed motion analysis system (Vicon, Oxford, England) sampling at 200 Hz will be used to record gait kinematics. The indicated anatomical landmarks (either C7 and T10 or posterior calcaneus and 2nd metatarsal phalangeal joint) will be marked with an ultraviolet pen, which will allow for visibility for a week, and will be reapplied at subsequent visits. This will improve marker placement repeatability during the gait retraining phase. A five-minute dynamic warm-up will be provided prior to the commencement of each gait retraining session; participants will then walk with their individualized gait modification strategy for 20 minutes. Participants will be provided with haptic feedback in the same manner outlined during the individualization phase or will continue to walk without feedback. A fading feedback design will be implemented across sessions to gradually integrate task acquisition and transfer and to help facilitate the internalization of the learned skill. During the first 2 weeks, real-time biofeedback (RTB) will be delivered on every step. For the third and fourth week, RTB will be provided on the first 3 foot strikes by the experimental leg and withheld on the fourth indicating a 25% reduction. During the fifth and sixth week, feedback will be provided on alternating foot strikes reducing RTB frequency delivery to 50%. For the final two weeks of gait-retraining, no feedback will be provided on the first three steps but delivered on the fourth reducing RTB frequency to 25%.

Between gait retraining sessions, subjects will be instructed to practice their acquired gait strategy on their own outside of the laboratory session, which will occur in the absence of feedback. They will be instructed to practice at least 10 min per day and will be provided weekly activity logs to record time of day and amount practiced each day during the eight weeks of gait retraining. Practice logs will be submitted weekly. Over-ground gait analysis and 12 minutes of treadmill walking will be performed at week 4 (first post-test) and 9 (2nd post-test) over the course of the intervention to track skill acquisition. This testing will be the same as the baseline trials, however, participants will be instructed to walk using only their specific gait modification strategy. No feedback will be provided during any of the skill acquisition or retention tests. Follow-up testing will occur at one, three, and six months as well as one-year post-intervention to measure retention of prescribed gait modifications.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of knee osteoarthritis by a qualified health professional such as an orthopedic surgeon or physical therapist
* between the ages of 18 and 80
* able to walk unaided for a minimum of 20 minutes

Exclusion Criteria:

* body mass index greater than 35
* history of lower back, hip or, knee surgery within the last 2 years
* knee arthroscopy or pharmacological injection in the previous six months
* neurological, or musculoskeletal conditions affecting ambulation
* cognitive impairment that would inhibit motor learning
* use of gait aid, orthotic shoe inserts, or hinged knee brace

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Knee Adduction Moment from Baseline at 10-weeks | It will be assessed using biomechanical analysis at baseline and 10-weeks gait retraining intervention
  The knee adduction moment is a surrogate measure to evaluate knee joint loads.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Cortes, Principal Investigator — Associate Professor
Locations (1):
- Sports Medicine, Assessment, Research & Testing (SMART) Laboratory, Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen KD, Golightly YM. State of the evidence. Curr Opin Rheumatol. 2015 May;27(3):276-83. doi: 10.1097/BOR.0000000000000161. PMID 25775186
- [Background] Amin S, Luepongsak N, McGibbon CA, LaValley MP, Krebs DE, Felson DT. Knee adduction moment and development of chronic knee pain in elders. Arthritis Rheum. 2004 Jun 15;51(3):371-6. doi: 10.1002/art.20396. PMID 15188321
- [Background] Anderson DI, Magill RA, Sekiya H, Ryan G. Support for an explanation of the guidance effect in motor skill learning. J Mot Behav. 2005 May;37(3):231-8. doi: 10.3200/JMBR.37.3.231-238. PMID 15883120
- [Background] Andriacchi TP, Mundermann A. The role of ambulatory mechanics in the initiation and progression of knee osteoarthritis. Curr Opin Rheumatol. 2006 Sep;18(5):514-8. doi: 10.1097/01.bor.0000240365.16842.4e. PMID 16896293
- [Background] Andriacchi TP, Mundermann A, Smith RL, Alexander EJ, Dyrby CO, Koo S. A framework for the in vivo pathomechanics of osteoarthritis at the knee. Ann Biomed Eng. 2004 Mar;32(3):447-57. doi: 10.1023/b:abme.0000017541.82498.37. PMID 15095819
- [Background] Barrios JA, Crossley KM, Davis IS. Gait retraining to reduce the knee adduction moment through real-time visual feedback of dynamic knee alignment. J Biomech. 2010 Aug 10;43(11):2208-13. doi: 10.1016/j.jbiomech.2010.03.040. Epub 2010 May 8. PMID 20452595
- [Background] Bellamy N, Buchanan WW. A preliminary evaluation of the dimensionality and clinical importance of pain and disability in osteoarthritis of the hip and knee. Clin Rheumatol. 1986 Jun;5(2):231-41. doi: 10.1007/BF02032362. PMID 3731718
- [Background] Bennell KL, Bowles KA, Wang Y, Cicuttini F, Davies-Tuck M, Hinman RS. Higher dynamic medial knee load predicts greater cartilage loss over 12 months in medial knee osteoarthritis. Ann Rheum Dis. 2011 Oct;70(10):1770-4. doi: 10.1136/ard.2010.147082. Epub 2011 Jul 7. PMID 21742637
- [Background] Bernier PM, Chua R, Franks IM. Is proprioception calibrated during visually guided movements? Exp Brain Res. 2005 Nov;167(2):292-6. doi: 10.1007/s00221-005-0063-5. Epub 2005 Nov 15. PMID 16044301
- [Background] Birmingham TB, Hunt MA, Jones IC, Jenkyn TR, Giffin JR. Test-retest reliability of the peak knee adduction moment during walking in patients with medial compartment knee osteoarthritis. Arthritis Rheum. 2007 Aug 15;57(6):1012-7. doi: 10.1002/art.22899. PMID 17665490
- [Background] Butler RJ, Minick KI, Ferber R, Underwood F. Gait mechanics after ACL reconstruction: implications for the early onset of knee osteoarthritis. Br J Sports Med. 2009 May;43(5):366-70. doi: 10.1136/bjsm.2008.052522. Epub 2008 Nov 28. PMID 19042923
- [Background] Chang AH, Moisio KC, Chmiel JS, Eckstein F, Guermazi A, Prasad PV, Zhang Y, Almagor O, Belisle L, Hayes K, Sharma L. External knee adduction and flexion moments during gait and medial tibiofemoral disease progression in knee osteoarthritis. Osteoarthritis Cartilage. 2015 Jul;23(7):1099-106. doi: 10.1016/j.joca.2015.02.005. Epub 2015 Feb 10. PMID 25677110
- [Background] Chang A, Hurwitz D, Dunlop D, Song J, Cahue S, Hayes K, Sharma L. The relationship between toe-out angle during gait and progression of medial tibiofemoral osteoarthritis. Ann Rheum Dis. 2007 Oct;66(10):1271-5. doi: 10.1136/ard.2006.062927. Epub 2007 Jan 31. PMID 17267516
- [Background] Chang JY, Chang GL, Chien CJ, Chung KC, Hsu AT. Effectiveness of two forms of feedback on training of a joint mobilization skill by using a joint translation simulator. Phys Ther. 2007 Apr;87(4):418-30. doi: 10.2522/ptj.20060154. Epub 2007 Mar 6. PMID 17341511
- [Background] Chehab EF, Favre J, Erhart-Hledik JC, Andriacchi TP. Baseline knee adduction and flexion moments during walking are both associated with 5 year cartilage changes in patients with medial knee osteoarthritis. Osteoarthritis Cartilage. 2014 Nov;22(11):1833-9. doi: 10.1016/j.joca.2014.08.009. Epub 2014 Aug 27. PMID 25211281
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of doctor-diagnosed arthritis and arthritis-attributable activity limitation--United States, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):869-73. PMID 24196662
- [Background] Zalecki T, Gorecka-Mazur A, Pietraszko W, Surowka AD, Novak P, Moskala M, Krygowska-Wajs A. Visual feedback training using WII Fit improves balance in Parkinson's disease. Folia Med Cracov. 2013;53(1):65-78. PMID 24858332
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Dearborn JT, Eakin CL, Skinner HB. Medial compartment arthrosis of the knee. Am J Orthop (Belle Mead NJ). 1996 Jan;25(1):18-26. PMID 8722125
- [Background] Deshpande BR, Katz JN, Solomon DH, Yelin EH, Hunter DJ, Messier SP, Suter LG, Losina E. Number of Persons With Symptomatic Knee Osteoarthritis in the US: Impact of Race and Ethnicity, Age, Sex, and Obesity. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1743-1750. doi: 10.1002/acr.22897. Epub 2016 Nov 3. PMID 27014966
- [Background] Dowling AV, Fisher DS, Andriacchi TP. Gait modification via verbal instruction and an active feedback system to reduce peak knee adduction moment. J Biomech Eng. 2010 Jul;132(7):071007. doi: 10.1115/1.4001584. PMID 20590285
- [Background] Duncan R, Peat G, Thomas E, Wood L, Hay E, Croft P. Does isolated patellofemoral osteoarthritis matter? Osteoarthritis Cartilage. 2009 Sep;17(9):1151-5. doi: 10.1016/j.joca.2009.03.016. Epub 2009 Apr 17. PMID 19401244
- [Background] Eddo, O., Lindsey, B., Caswell, S. V., & Cortes, N. (2017). Current Evidence of Gait Modification with Real-time Biofeedback to Alter Kinetic, Temporospatial, and Function-Related Outcomes: A Review. International Journal of Kinesiology and Sports Science, 5(3), 35-55.
- [Background] Favre J, Erhart-Hledik JC, Chehab EF, Andriacchi TP. General scheme to reduce the knee adduction moment by modifying a combination of gait variables. J Orthop Res. 2016 Sep;34(9):1547-56. doi: 10.1002/jor.23151. Epub 2016 Jan 21. PMID 26744298
- [Background] Felson DT. Clinical practice. Osteoarthritis of the knee. N Engl J Med. 2006 Feb 23;354(8):841-8. doi: 10.1056/NEJMcp051726. No abstract available. PMID 16495396
- [Background] Ferrigno C, Stoller IS, Shakoor N, Thorp LE, Wimmer MA. The Feasibility of Using Augmented Auditory Feedback From a Pressure Detecting Insole to Reduce the Knee Adduction Moment: A Proof of Concept Study. J Biomech Eng. 2016 Feb;138(2):021014. doi: 10.1115/1.4032123. PMID 26632644
- [Background] Foroughi N, Smith R, Vanwanseele B. The association of external knee adduction moment with biomechanical variables in osteoarthritis: a systematic review. Knee. 2009 Oct;16(5):303-9. doi: 10.1016/j.knee.2008.12.007. Epub 2009 Mar 24. PMID 19321348
- [Background] Fregly BJ, Reinbolt JA, Rooney KL, Mitchell KH, Chmielewski TL. Design of patient-specific gait modifications for knee osteoarthritis rehabilitation. IEEE Trans Biomed Eng. 2007 Sep;54(9):1687-95. doi: 10.1109/tbme.2007.891934. PMID 17867361
- [Background] Gerbrands TA, Pisters MF, Vanwanseele B. Individual selection of gait retraining strategies is essential to optimally reduce medial knee load during gait. Clin Biomech (Bristol). 2014 Aug;29(7):828-34. doi: 10.1016/j.clinbiomech.2014.05.005. Epub 2014 May 27. PMID 24917175
- [Background] Greska EK, Cortes N, Ringleb SI, Onate JA, Van Lunen BL. Biomechanical differences related to leg dominance were not found during a cutting task. Scand J Med Sci Sports. 2017 Nov;27(11):1328-1336. doi: 10.1111/sms.12776. Epub 2016 Oct 17. PMID 27747935
- [Background] Grood ES, Suntay WJ. A joint coordinate system for the clinical description of three-dimensional motions: application to the knee. J Biomech Eng. 1983 May;105(2):136-44. doi: 10.1115/1.3138397. PMID 6865355
- [Background] Heijink A, Gomoll AH, Madry H, Drobnic M, Filardo G, Espregueira-Mendes J, Van Dijk CN. Biomechanical considerations in the pathogenesis of osteoarthritis of the knee. Knee Surg Sports Traumatol Arthrosc. 2012 Mar;20(3):423-35. doi: 10.1007/s00167-011-1818-0. Epub 2011 Dec 16. PMID 22173730
- [Background] Hootman JM, Helmick CG, Barbour KE, Theis KA, Boring MA. Updated Projected Prevalence of Self-Reported Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation Among US Adults, 2015-2040. Arthritis Rheumatol. 2016 Jul;68(7):1582-7. doi: 10.1002/art.39692. PMID 27015600
- [Background] Hunt MA, Simic M, Hinman RS, Bennell KL, Wrigley TV. Feasibility of a gait retraining strategy for reducing knee joint loading: increased trunk lean guided by real-time biofeedback. J Biomech. 2011 Mar 15;44(5):943-7. doi: 10.1016/j.jbiomech.2010.11.027. Epub 2010 Dec 7. PMID 21144522
- [Background] Hunt MA, Takacs J. Effects of a 10-week toe-out gait modification intervention in people with medial knee osteoarthritis: a pilot, feasibility study. Osteoarthritis Cartilage. 2014 Jul;22(7):904-11. doi: 10.1016/j.joca.2014.04.007. Epub 2014 May 14. PMID 24836210
- [Background] Hunter DJ, March L, Sambrook PN. The association of cartilage volume with knee pain. Osteoarthritis Cartilage. 2003 Oct;11(10):725-9. doi: 10.1016/s1063-4584(03)00160-2. PMID 13129691
- [Background] Hurwitz DE, Ryals AB, Case JP, Block JA, Andriacchi TP. The knee adduction moment during gait in subjects with knee osteoarthritis is more closely correlated with static alignment than radiographic disease severity, toe out angle and pain. J Orthop Res. 2002 Jan;20(1):101-7. doi: 10.1016/S0736-0266(01)00081-X. PMID 11853076
- [Background] Jackson BD, Wluka AE, Teichtahl AJ, Morris ME, Cicuttini FM. Reviewing knee osteoarthritis--a biomechanical perspective. J Sci Med Sport. 2004 Sep;7(3):347-57. doi: 10.1016/s1440-2440(04)80030-6. PMID 15518300
- [Background] Kaufman KR, Hughes C, Morrey BF, Morrey M, An KN. Gait characteristics of patients with knee osteoarthritis. J Biomech. 2001 Jul;34(7):907-15. doi: 10.1016/s0021-9290(01)00036-7. PMID 11410174
- [Background] Kean CO, Bennell KL, Wrigley TV, Hinman RS. Modified walking shoes for knee osteoarthritis: Mechanisms for reductions in the knee adduction moment. J Biomech. 2013 Aug 9;46(12):2060-6. doi: 10.1016/j.jbiomech.2013.05.011. Epub 2013 Jun 14. PMID 23768609
- [Background] Kean CO, Hinman RS, Bowles KA, Cicuttini F, Davies-Tuck M, Bennell KL. Comparison of peak knee adduction moment and knee adduction moment impulse in distinguishing between severities of knee osteoarthritis. Clin Biomech (Bristol). 2012 Jun;27(5):520-3. doi: 10.1016/j.clinbiomech.2011.12.007. Epub 2012 Jan 12. PMID 22244512
- [Background] Kumar D, Manal KT, Rudolph KS. Knee joint loading during gait in healthy controls and individuals with knee osteoarthritis. Osteoarthritis Cartilage. 2013 Feb;21(2):298-305. doi: 10.1016/j.joca.2012.11.008. Epub 2012 Nov 24. PMID 23182814
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839
- [Background] Maly MR, Robbins SM, Stratford PW, Birmingham TB, Callaghan JP. Cumulative knee adductor load distinguishes between healthy and osteoarthritic knees--a proof of principle study. Gait Posture. 2013 Mar;37(3):397-401. doi: 10.1016/j.gaitpost.2012.08.013. Epub 2012 Sep 18. PMID 22995753
- [Background] Manal K, Gardinier E, Buchanan TS, Snyder-Mackler L. A more informed evaluation of medial compartment loading: the combined use of the knee adduction and flexor moments. Osteoarthritis Cartilage. 2015 Jul;23(7):1107-11. doi: 10.1016/j.joca.2015.02.779. Epub 2015 Apr 8. PMID 25862486
- [Background] Mandelbaum B, Waddell D. Etiology and pathophysiology of osteoarthritis. Orthopedics. 2005 Feb;28(2 Suppl):s207-14. doi: 10.3928/0147-7447-20050202-05. PMID 15747608
- [Background] Mayr A, Kofler M, Quirbach E, Matzak H, Frohlich K, Saltuari L. Prospective, blinded, randomized crossover study of gait rehabilitation in stroke patients using the Lokomat gait orthosis. Neurorehabil Neural Repair. 2007 Jul-Aug;21(4):307-14. doi: 10.1177/1545968307300697. Epub 2007 May 2. PMID 17476001
- [Background] Miyazaki T, Wada M, Kawahara H, Sato M, Baba H, Shimada S. Dynamic load at baseline can predict radiographic disease progression in medial compartment knee osteoarthritis. Ann Rheum Dis. 2002 Jul;61(7):617-22. doi: 10.1136/ard.61.7.617. PMID 12079903
- [Background] Mundermann A, Asay JL, Mundermann L, Andriacchi TP. Implications of increased medio-lateral trunk sway for ambulatory mechanics. J Biomech. 2008;41(1):165-70. doi: 10.1016/j.jbiomech.2007.07.001. Epub 2007 Aug 3. PMID 17678933
- [Background] Mundermann A, Dyrby CO, Andriacchi TP. Secondary gait changes in patients with medial compartment knee osteoarthritis: increased load at the ankle, knee, and hip during walking. Arthritis Rheum. 2005 Sep;52(9):2835-44. doi: 10.1002/art.21262. PMID 16145666
- [Background] Murphy DF, Connolly DA, Beynnon BD. Risk factors for lower extremity injury: a review of the literature. Br J Sports Med. 2003 Feb;37(1):13-29. doi: 10.1136/bjsm.37.1.13. PMID 12547739
- [Background] Murphy LB, Cisternas MG, Pasta DJ, Helmick CG, Yelin EH. Medical Expenditures and Earnings Losses Among US Adults With Arthritis in 2013. Arthritis Care Res (Hoboken). 2018 Jun;70(6):869-876. doi: 10.1002/acr.23425. Epub 2018 Apr 16. PMID 28950426
- [Background] Neogi T, Zhang Y. Epidemiology of osteoarthritis. Rheum Dis Clin North Am. 2013 Feb;39(1):1-19. doi: 10.1016/j.rdc.2012.10.004. Epub 2012 Nov 10. PMID 23312408
- [Background] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Background] Noehren B, Scholz J, Davis I. The effect of real-time gait retraining on hip kinematics, pain and function in subjects with patellofemoral pain syndrome. Br J Sports Med. 2011 Jul;45(9):691-6. doi: 10.1136/bjsm.2009.069112. Epub 2010 Jun 28. PMID 20584755
- [Background] Richards RE, Andersen MS, Harlaar J, van den Noort JC. Relationship between knee joint contact forces and external knee joint moments in patients with medial knee osteoarthritis: effects of gait modifications. Osteoarthritis Cartilage. 2018 Sep;26(9):1203-1214. doi: 10.1016/j.joca.2018.04.011. Epub 2018 Apr 30. PMID 29715509
- [Background] Richards R, van den Noort JC, van der Esch M, Booij MJ, Harlaar J. Gait retraining using real-time feedback in patients with medial knee osteoarthritis: Feasibility and effects of a six-week gait training program. Knee. 2018 Oct;25(5):814-824. doi: 10.1016/j.knee.2018.05.014. Epub 2018 Jun 20. PMID 29933935
- [Background] Richards RE, van den Noort JC, van der Esch M, Booij MJ, Harlaar J. Effect of real-time biofeedback on peak knee adduction moment in patients with medial knee osteoarthritis: Is direct feedback effective? Clin Biomech (Bristol). 2018 Aug;57:150-158. doi: 10.1016/j.clinbiomech.2017.07.004. Epub 2017 Jul 13. PMID 28811046
- [Background] Richards R, van den Noort JC, Dekker J, Harlaar J. Gait Retraining With Real-Time Biofeedback to Reduce Knee Adduction Moment: Systematic Review of Effects and Methods Used. Arch Phys Med Rehabil. 2017 Jan;98(1):137-150. doi: 10.1016/j.apmr.2016.07.006. Epub 2016 Jul 30. PMID 27485366
- [Background] Riskowski JL. Gait and neuromuscular adaptations after using a feedback-based gait monitoring knee brace. Gait Posture. 2010 Jun;32(2):242-7. doi: 10.1016/j.gaitpost.2010.05.002. Epub 2010 Jun 16. PMID 20558068
- [Background] Schwartz MH, Rozumalski A. A new method for estimating joint parameters from motion data. J Biomech. 2005 Jan;38(1):107-16. doi: 10.1016/j.jbiomech.2004.03.009. PMID 15519345
- [Background] Segal NA, Glass NA, Teran-Yengle P, Singh B, Wallace RB, Yack HJ. Intensive Gait Training for Older Adults with Symptomatic Knee Osteoarthritis. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):848-58. doi: 10.1097/PHM.0000000000000264. PMID 25768068
- [Background] Sharma L, Lou C, Cahue S, Dunlop DD. The mechanism of the effect of obesity in knee osteoarthritis: the mediating role of malalignment. Arthritis Rheum. 2000 Mar;43(3):568-75. doi: 10.1002/1529-0131(200003)43:33.0.CO;2-E. PMID 10728750
- [Background] Sharma L, Hurwitz DE, Thonar EJ, Sum JA, Lenz ME, Dunlop DD, Schnitzer TJ, Kirwan-Mellis G, Andriacchi TP. Knee adduction moment, serum hyaluronan level, and disease severity in medial tibiofemoral osteoarthritis. Arthritis Rheum. 1998 Jul;41(7):1233-40. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-L. PMID 9663481
- [Background] Shull, P., Lurie, K., Shin, M., Besier, T., & Cutkosky, M. (2010). Haptic gait retraining for knee osteoarthritis treatment. In 2010 IEEE Haptics Symposium (pp. 409-416)
- [Background] Shull PB, Lurie KL, Cutkosky MR, Besier TF. Training multi-parameter gaits to reduce the knee adduction moment with data-driven models and haptic feedback. J Biomech. 2011 May 17;44(8):1605-9. doi: 10.1016/j.jbiomech.2011.03.016. Epub 2011 Apr 2. PMID 21459384
- [Background] Shull PB, Shultz R, Silder A, Dragoo JL, Besier TF, Cutkosky MR, Delp SL. Toe-in gait reduces the first peak knee adduction moment in patients with medial compartment knee osteoarthritis. J Biomech. 2013 Jan 4;46(1):122-8. doi: 10.1016/j.jbiomech.2012.10.019. Epub 2012 Nov 10. PMID 23146322
- [Background] Shull PB, Silder A, Shultz R, Dragoo JL, Besier TF, Delp SL, Cutkosky MR. Six-week gait retraining program reduces knee adduction moment, reduces pain, and improves function for individuals with medial compartment knee osteoarthritis. J Orthop Res. 2013 Jul;31(7):1020-5. doi: 10.1002/jor.22340. Epub 2013 Mar 12. PMID 23494804
- [Background] Shull PB, Damian DD. Haptic wearables as sensory replacement, sensory augmentation and trainer - a review. J Neuroeng Rehabil. 2015 Jul 20;12:59. doi: 10.1186/s12984-015-0055-z. PMID 26188929
- [Background] Sigrist R, Rauter G, Riener R, Wolf P. Augmented visual, auditory, haptic, and multimodal feedback in motor learning: a review. Psychon Bull Rev. 2013 Feb;20(1):21-53. doi: 10.3758/s13423-012-0333-8. PMID 23132605
- [Background] Silverwood V, Blagojevic-Bucknall M, Jinks C, Jordan JL, Protheroe J, Jordan KP. Current evidence on risk factors for knee osteoarthritis in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Apr;23(4):507-15. doi: 10.1016/j.joca.2014.11.019. Epub 2014 Nov 29. PMID 25447976
- [Background] Simic M, Wrigley TV, Hinman RS, Hunt MA, Bennell KL. Altering foot progression angle in people with medial knee osteoarthritis: the effects of varying toe-in and toe-out angles are mediated by pain and malalignment. Osteoarthritis Cartilage. 2013 Sep;21(9):1272-80. doi: 10.1016/j.joca.2013.06.001. PMID 23973141
- [Background] Simic M, Hinman RS, Wrigley TV, Bennell KL, Hunt MA. Gait modification strategies for altering medial knee joint load: a systematic review. Arthritis Care Res (Hoboken). 2011 Mar;63(3):405-26. doi: 10.1002/acr.20380. Epub 2010 Oct 27. PMID 20981808
- [Background] Simic M, Hunt MA, Bennell KL, Hinman RS, Wrigley TV. Trunk lean gait modification and knee joint load in people with medial knee osteoarthritis: the effect of varying trunk lean angles. Arthritis Care Res (Hoboken). 2012 Oct;64(10):1545-53. doi: 10.1002/acr.21724. PMID 22556125
- [Background] Simon D, Mascarenhas R, Saltzman BM, Rollins M, Bach BR Jr, MacDonald P. The Relationship between Anterior Cruciate Ligament Injury and Osteoarthritis of the Knee. Adv Orthop. 2015;2015:928301. doi: 10.1155/2015/928301. Epub 2015 Apr 19. PMID 25954533
- [Background] Snodgrass SJ, Rivett DA, Robertson VJ, Stojanovski E. Real-time feedback improves accuracy of manually applied forces during cervical spine mobilisation. Man Ther. 2010 Feb;15(1):19-25. doi: 10.1016/j.math.2009.05.011. Epub 2009 Jul 25. PMID 19632877
- [Background] Sulzenbruck S, Heuer H. Type of visual feedback during practice influences the precision of the acquired internal model of a complex visuo-motor transformation. Ergonomics. 2011 Jan;54(1):34-46. doi: 10.1080/00140139.2010.535023. PMID 21181587
- [Background] Tate JJ, Milner CE. Real-time kinematic, temporospatial, and kinetic biofeedback during gait retraining in patients: a systematic review. Phys Ther. 2010 Aug;90(8):1123-34. doi: 10.2522/ptj.20080281. Epub 2010 Jun 17. PMID 20558567
- [Background] Teng HL, MacLeod TD, Link TM, Majumdar S, Souza RB. Higher Knee Flexion Moment During the Second Half of the Stance Phase of Gait Is Associated With the Progression of Osteoarthritis of the Patellofemoral Joint on Magnetic Resonance Imaging. J Orthop Sports Phys Ther. 2015 Sep;45(9):656-64. doi: 10.2519/jospt.2015.5859. Epub 2015 Jul 10. PMID 26161626
- [Background] Thomas RH, Resnick D, Alazraki NP, Daniel D, Greenfield R. Compartmental evaluation of osteoarthritis of the knee. A comparative study of available diagnostic modalities. Radiology. 1975 Sep;116(3):585-94. doi: 10.1148/116.3.585. PMID 1153764
- [Background] Thorp LE, Sumner DR, Block JA, Moisio KC, Shott S, Wimmer MA. Knee joint loading differs in individuals with mild compared with moderate medial knee osteoarthritis. Arthritis Rheum. 2006 Dec;54(12):3842-9. doi: 10.1002/art.22247. PMID 17133592
- [Background] Uhlrich SD, Silder A, Beaupre GS, Shull PB, Delp SL. Subject-specific toe-in or toe-out gait modifications reduce the larger knee adduction moment peak more than a non-personalized approach. J Biomech. 2018 Jan 3;66:103-110. doi: 10.1016/j.jbiomech.2017.11.003. Epub 2017 Nov 8. PMID 29174534
- [Background] van den Noort JC, Steenbrink F, Roeles S, Harlaar J. Real-time visual feedback for gait retraining: toward application in knee osteoarthritis. Med Biol Eng Comput. 2015 Mar;53(3):275-86. doi: 10.1007/s11517-014-1233-z. Epub 2014 Dec 6. PMID 25480419
- [Background] Walter JP, D'Lima DD, Colwell CW Jr, Fregly BJ. Decreased knee adduction moment does not guarantee decreased medial contact force during gait. J Orthop Res. 2010 Oct;28(10):1348-54. doi: 10.1002/jor.21142. PMID 20839320
- [Background] Wheeler JW, Shull PB, Besier TF. Real-time knee adduction moment feedback for gait retraining through visual and tactile displays. J Biomech Eng. 2011 Apr;133(4):041007. doi: 10.1115/1.4003621. PMID 21428681
- [Background] Winstein CJ. Knowledge of results and motor learning--implications for physical therapy. Phys Ther. 1991 Feb;71(2):140-9. doi: 10.1093/ptj/71.2.140. PMID 1989009
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Zhao D, Banks SA, Mitchell KH, D'Lima DD, Colwell CW Jr, Fregly BJ. Correlation between the knee adduction torque and medial contact force for a variety of gait patterns. J Orthop Res. 2007 Jun;25(6):789-97. doi: 10.1002/jor.20379. PMID 17343285